CLINICAL TRIAL: NCT06499103
Title: Effects of Transcutaneous Electrical Nerve Stimulation on Chemotherapy-induced Peripheral Neuropathy Symptoms
Brief Title: Effect of Transcutaneous Electrical Nerve Stimulation on CIPN Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jordan University of Science and Technology (Other)
Collaborators: King hussein cancer foundation and center (Unknown)
Responsible Party: Principal Investigator, Nour Alazam, Principal Investigator, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TENS on CIPN
Record Dates: First submitted 2022-10-26; First posted 2024-07-12 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Cancer; Chemotherapy; Transcutaneous electrical nerve stimulation; Chemotherapy-induced peripheral neuropathy
MeSH Terms: conditions — Neoplasms | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): The interventional group (n=22) will receive TENS sessions in addition to the prescribes medication (Gabapentinoids). The assessment will be performed at three time points also; before the begging of the intervention, after 5 days, and after the last session.
  Interventions: Device: Transcutaneous electrical nerve stimulation
- Control group (No Intervention): The control group The control group (n=22) will stay on the prescribed oral medication (Gabapentinoids) for at least 4 weeks (Hirayama et al.,2015). The assessment will be performed at three time points by the primary investigator using the Arabic version of CIPNAT . The first assessment will take place prior to the start of the trial, after two weeks of taking the medication, and the final assessment will be done after 4 weeks of receiving oral agents.

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation — The stimulation (TENS) will be performed by a physiotherapist using adhesive electrodes with an area of 5 cm2 in the region where the patient has the symptoms of neuropathy. Further, it will be will be on 10 days consequently, with the same physiotherapist for whole sessions. He will apply electrodes over the affected area, then he will increase the stimulation intensity gradually during the first session when he adjusts the settings till patient reach the maximum voltage that he/she will tolerate it. The evaluations for CIPN patients will be performed by a blinded evaluatorthe PI on the experimental groups at 3 time points; before the begging of the intervention, after 5 days, and after the last session. The intervention group will undergo TENS sessions daily for 10 days for 30 minutes each session ( Gibson et al., 2017). After session completed a structured interview will be conducted, by the primary investigator, to assess for CIPN using the CIPNAT.
  Arms: Interventional group

SUMMARY:
Background: Chemotherapy-induced peripheral neuropathy (CIPN) is one of the most common and debilitating survivorship conditions for patients with cancer, and one of the most common side effects of chemotherapy treatment. Unfortunately, there are no proven ways to prevent or treat CIPN. Transcutaneous electrical nerve stimulation (TENS) is a method that succeeded to treat different types of pain and needs more investigation on its effect on CIPN.

Aim : The aims of this study are to investigate the effect of TENS in reducing CIPN symptoms in patients with cancer and to investigate the relathionship between some of the patients' sociodemographic charestristics/ medical history and the levels of CIPN after treatment with TENS.

Method : A double blind parallel randomized controlled trial (RCT) will be used in this study to assess the effect of TENS on CIPN among patients with cancer treated with chemotherapy. Participants will be recruited from King Hussein Cancer Center (KHCC). 44 patients will be included in the study if they developed CIPN after the first cycle of chemotherapy treatment, were ≥18 years old, and were not previously received any session of TENS device and only on gabapentin drug currently. Patients will be randomly assigned to one of two groups, 22 patient for each group. The intervention group will receive the TENS sessions daily for 10 days and for 30 minutes each session. The control group will stay on gabapentin. CIPN will be assessed using the Arabic Version of the Chemotherapy-Induced Peripheral Neuropathy Assessment Tool. CIPN will be assessed three time during the study: first time will be pre-intervention, second time will be after 5 days of treatment and the third time will be at the end of the sessions.

Implication : The result will lead nursing to achieve optimal nursing care for all patients by controlling the pain level and improve other peripheral neuropathy symptoms .

DETAILED DESCRIPTION:
Chemotherapy Induced Peripheral Neuropathy (CIPN) is a common and serious side effect of chemotherapy treatment that causes autonomic neurons, sensory, or motor nerve damage or dysfunction. CIPN develop in some patients gradually over months to years, while in others may develop rapidly and continue to get worse during or immediately after infusion.

It was found that CIPN can also affected by race and gender. African American women exhibited two to three times higher risk for developing CIPN relative to White Women Further, non-Chinese Asians had a higher risk of developing neuropathy than Chinese or Caucasians in One study (n=255) investigated patients receiving platinum- and taxane based chemotherapy for a variety of solid tumors in Hong Kong, Singapore.

Thus, CIPN need to be managed and solved to prevent CIPN before it occurs and to alleviate symptoms after CIPN has developed. In terms of prophylaxis, American Society of Clinical Oncology (ASCO) practice recommendations state that there is no proven way to prevent, mitigate, or manage CIPN occurrence. Despite trials indicating modest effectiveness, many practitioners explore the use of neuropathic pain medications such as gabapentin, pregabalin, tricyclic antidepressants, and others for symptomatic relief. Nevertheless, only venlafaxine and duloxetine have been shown to be effective in alleviation paresthesia. Duloxetine (orally) is currently the only FDA-approved medication for the treatment of established CIPN and is an ASCO recommended therapy for patients.

Alternative and complementary medicine methods to treat CIPN have also been studied. Firstly, acupuncture is one such technique that is becoming more popular as an effective supplement to other treatments for CIPN. Secondly, Neuromodulation involves electrical stimulation of peripheral nerves (e.g., transcutaneous electrical nerve stimulators, Scrambler therapy) or modulation of the central processing of painful afferent impulses via real-time feedback using electroencephalography to "retrain" the brain to perceive neuropathic pain as a nonpainful stimulus (e.g. neurofeedback). Thirdly, scrambler treatment for CIPN has mainly favorable results, although heterogeneity and small sample sizes restrict it. Fourthly, exercise and cannabinoids are two treatments for CIPN that have a growing body of clinical and preclinical data to back them up.

Transcutaneous Electrical Nerve Stimulation (TENS) has considered as an alternative treatment to conventional pharmacotherapy for cancer patients having CIPN. TENS machine is a non-invasive, inexpensive therapy, operated by a battery. It activates peripheral nerves by delivering low-voltage electrical impulses to control any type of pain (localized, acute or chronic) through 2 -4 sticky electrodes connect via wires placed on the surface of skin, which could blocks or changes the perception of pain.

TENS has shown a positive effect on nerve regeneration, axon density, revealing a higher number of myelinated fibers, and blood vessels in the nerve area. Further, the electrical stimulation could enhance and raise regeneration and rehabilitation interventions to improve sensorimotor skills after peripheral nerve injury.

TENS is an FDA approved therapy that commonly used to treat a variety of neuropathic pain. It was applied successfully to treat some surgeries as oral-facial surgeries, and labor pain, diabetic peripheral neuropathy, fibromyalgia, and migraine.

TENS device does not decrease the pain level and neuropathic symptoms only, it can increase blood circulation, stimulates skin wound healing and tendon repair (Machado et al., 2012), decreases inflammation.

However, few research have been done on the effect of TENS on CIPN. Therefore, this study is aimed to investigate the effect of TENS on CIPN among cancer patients.

Statement of the Problem:

Approximately 50-90% of patients who are treated with chemotherapy are affected by CIPN and bear a high risk of chronicity. According to a meta-analysis, the aggregate prevalence of CIPN is estimated to be 48%. The prevalence of CIPN is expected to increase in the future if new treatment protocols use more intensive dosing or combinations of neurotoxic chemotherapy agents or if cancer patients who were treated with neurotoxic chemotherapy experience prolonged survival.

Although clinical trials evaluating CIPN prevention or treatment have generally failed to bring effective treatments into the clinic, some of the prophylactic and treating medications provide modest improvements in neurological function. However, in most instances, these agents are associated with additional negative side effects for cancer patients including cardiac conduction defects and increased chemotherapy resistance, which affect the patients' quality of life (QoL).

As a result of that, health care providers may reduce the does or discontinue the chemotherapeutic drugs to limit the severity of CIPN. That could result in treatment delay, and possibly negative impact on the cancer treatment, disease control and progress and alleviate symptoms of CIPN .

According to the American Cancer Society, CIPN is an under-addressed problem in oncology and little attention has been given to the deleterious effects of CIPN. With CIPN becoming a growing problem, new methods of treating CIPN and its negative influence on physical performance must be discovered. TENS is an innovative and FDA approved method in Jordan to treat a variety of neuropathic pain. It has documented effects in reducing pain related to different pathologies as well as CIPN. However, few studies addressed the effect of TENS on reducing CIPN among cancer patients. Further, there is no studies discussed this subject in Jordan. Therefore, the purpose of this study is to investigate the effect of TENS in reducing CIPN symptoms among cancer patients.

Significant of the study: This study will be the first study to investigate the effect of TENS on the CIPN in Jordan as well as one of few studies around the world. Thus, it will add important information to the literature regarding the effect of TENS on CIPN. Further, it will spotlight on the effectiveness of TENS on the treatment of CIPN compared to the medications that cause serious side effects, and this strongly supports the need to develop future high quality, sufficiently powered trials. Moreover, health care providers including nurses would be able to weigh the risks and benefits of TENS compared to the medication in the treatment of CIPN and can direct the patients to the appropriate treatment. Therefore, the development of safe and effective interventions to prevent, mitigate or manage CIPN would represent an important medical advancement for patients with cancer.

Symptom management is the primary focus of oncology nursing. CIPN is an unpleasant symptom that can potentially adversely affect the quality of life (QOL), function, and safety of patients with cancer. Nurses can advocate on behalf of patients by understanding the distressing influence and long-term sequella CIPN can have on daily living. Nurses have a crucial role in providing symptom management to oncology patients. Therefore, lower level of pain, would increase patients' satisfaction with nursing care, which is one of our nursing goals and commonly used indicators for measuring the quality of health care. Further, symptoms management are multidisciplinary approach. nurse, physician, pharmacist, and physiotherapist assist each other's in managing symptoms.

This study will determine a non-pharmacological treatment for CIPN symptoms management. So, if TENS has a strong relationship with neuropathy symptoms and function, it could be used to avoid exposing the patient to medication and to guide clinicians to continue treatment protocol and avoid change the type, and dose reduction, or discontinuation of the neurotoxic chemotherapy. Further, it will help nurses and other health care professionals design and implement interventions to help prevent symptoms, recognize symptoms earlier, and treat symptoms more effectively.

Methodology: Design: A double blind parallel randomized controlled trial (RCT) will be used in this study to assess the effect of TENS on CIPN among patients with cancer treated with chemotherapy. RCT is a gold standard method that allows to infer causal relationship.

Sample and Setting:

A Random sample of patients with cancer will be recruited from King Hussein Cancer Center (KHCC), which is a specialized setting, providing comprehensive cancer care in Jordan. This center receives cancer cases from all over the Hashemite Kingdom of Jordan and the region. The outpatient chemotherapy clinics serve about 100 patients on a daily bases.

patients will be invited to participate in the study if they developed CIPN after the first cycle of chemotherapy treatment of grade I or grade II on the Common Terminology Criteria for Adverse Events (CTCAE) scale, with at least two points on the visual analog scale of paresthesia and/or pain, and having a present performance status of ECOG ≤2 (Karnofsky≥50%). Further, patients will be invited if they ≥18 years old, and were not previously received any session of TENS device and only on gabapentin drug currently. Patients will be excluded from the study if they have any skin conditions, such as lesions or open sores where the electrodes need to be placed, cognitive difficulties or trouble understanding how to fill out questionnaire, history of peripheral neuropathy due to receiving neurotoxic chemotherapy, cardiac pacemakers, or if they used TENS device treatment previously. Further, patients who have chronic conditions such as diabetes mellitus, brain damage, history of epilepsy, or taking anticonvulsants drugs as well as pregnant women will be excluded from the study.

Appropriate sample size will be calculated by performing the G-Power analysis using A-priori Sample Size Calculator for F-test. Given an alpha level of 0.05, an anticipated effect size of 0.25, the desired statistical power level of 0.8, number of groups 2, number of measurements 3, the minimum required sample size is 44 subjects, 22 subject for each group.

CIPN will be assessed using the Arabic Version of the Chemotherapy-Induced Peripheral Neuropathy Assessment Tool (CIPNAT). The original CIPNAT was developed by Tofthagen et al. (2011) based on the theory of Unpleasant Symptoms that suggests that complete assessment of unpleasant symptoms should include evaluation of symptom occurrence, severity, distress, frequency, and interference with daily activities. The original version of the CIPNAT consisted of 50 items. The CIPNAT has two assessment scales: One is the symptom assessment scale, and the other is the interference with activity scale.

The symptom experience scale has 36 items evaluate nine neuropathy symptoms with their characteristics (occurrence, severity, distress, and frequency). The patients indicate whether each symptom is present by answering a yes/no question and if yes, the symptom description items are answered on 0-10 Likert scales. The total possible score from each symptom is 31. This scale is scored from 0-279, which reflects the symptoms experienced in nine questions (0-1 for nine yes-or-no questions and 0-10 for the three sub-questions "severity," "distress," and "frequency"). With zero being no symptom and 10 being the worst possible. Cronbach alpha was (alpha = .93).

The interference with activity scale has 14 items including walking, picking up objects, holding into objects, driving, working, participating in hobbies or leisure activities, exercising, sexual activity, sleeping, relationships, writing, usual household chores, and enjoyment of life. Each item is scored from 0-10. This scale gives scores from 0-140 for the 14 items. Higher scores indicate increased severity of symptoms. Construct validity was tested for the interference with activity scale (t=4.81, p< .001). Internal consistency was demonstrated using Cronbach's alpha (alpha = .91).

Answering the first four questions indicates the presence or absence of chemotherapy-induced peripheral neuropathy. If the answer is "no" for the first four questions, the patient may stop and does not need to complete the rest of the questions due to absence of chemotherapy-induced peripheral neuropathy.

CIPNAT is shown to be sufficiently reliable and valid for screening for chemotherapy-induced peripheral neuropathy symptoms and their impairment with their interference daily activities in Arab countries. Validity and reliability of the total CIPNAT were tested by administering it to two groups of patients. One group had neuropathy, and the other did not. Content validity index generated by a panel of experts was acceptable at 0.95. Convergent validity data were provided by correlation with the Functional Assessment of Cancer Therapy/Gynecologic Oncology Group Neurotoxicity Scale (FACT/GOG-Ntx) (r = 0.83, P < .001) and differences between the compared groups (t = 7.66, P < .001) provided evidence of discriminant validity. High test-retest correlations (r = 0.92, P < .001), Cronbach's alpha = .95 and significant item-to-total correlations ranging from 0.38 to 0.70 provided evidence of reliability..

The Arabic version of CIPNAT contains 48 items that measure CIPN. The items ask about the characteristics, intensity, frequency, distress, and interference of CIPN with usual activities, such as changing clothes (buttoning a shirt, pulling the zipper of pants ... etc.), walking, picking up objects, driving, working, participating in hobbies or leisure activities, sleeping, sexual activity, relationships, writing, usual household chores, enjoyment of life. The maximum possible score is 10 which represent a sever CIPN symptoms intensity and the minimum score is zero which represent no CIPN symptoms based on Numerical rating scales (NRS). For the NRS, it is ordinal scale. Test-retest reliability evaluation was performed to evaluate the reliability of the Arabic version of CIPNAT.

Discriminant validity testing-the known-groups technique-was used. The instrument was administered on two groups of patients with cancer: patients who received chemotherapeutic agents with a high probability of causing CIPN symptoms versus patients who received chemotherapeutic agents with a low risk of causing neuropathic symptoms. Whereas, the content validity was evaluated by five experts, who evaluated whether the items accurately represented the characteristics of CIPN. The experts included a neurologist, medical oncologist, chemotherapy nurse, pain nurse, and pain physician. Experts were asked to assess every item in the tool to determine the extent of relevancy to chemotherapy-induced peripheral neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* patients will be invited if they ≥18 years
* were not previously received any session of TENS device
* on gabapentin drug currently

Exclusion Criteria:

* skin conditions (lesions or open sores)
* cognitive difficulties or trouble understanding
* history of peripheral neuropathy due to receiving neurotoxic chemotherapy
* cardiac pacemakers
* have ever used TENS device treatment
* chronic conditions (diabetes mellitus, brain damage, history of epilepsy, or taking anticonvulsants drugs)
* pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-08 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-06-29 (Actual)

PRIMARY OUTCOMES:
Effects of transcutaneous electrical nerve stimulation on chemotherapy-induced peripheral neuropathy symptoms: A randomized controlled trial | Baseline
  Participants scores in CTCAE and visual analog scales that measure the severity of adverse events of treatment and pain score.
  Retrospectively, showed improvement in both groups. However the interventional group (TENS with gabapentin) showed a higher reduction in total scores of scales compared with control group.

CONTACTS AND LOCATIONS:
Overall Officials: Nour Al-azzam, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan university of science and technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code